CLINICAL TRIAL: NCT04700943
Title: Ultrasound Assessment of Diaphragmatic Dysfunction: General Versus Regional Anesthesia for Video-assisted Thoracoscopic Surgery Pulmonary Biopsy in Interstitial Lung Disease
Brief Title: Ultrasound Assessment of Diaphragmatic Dysfunction in Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: DULORATHO
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Regional Anesthesia; Diaphragm Issues; Thoracic Surgery; Ultrasounds
Keywords: Ultrasounds; diaphragmatic function; thoracic surgery; regional anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regional awake anesthesia: In non-intubated patients, an epidural catheter was placed at T5-T6. An anesthetic load of 0,5 mg/kg of ropivacaine was administered to reach anesthesia of the thoracic wall. Adjunctive local anesthetic infiltration of the incision site was performed by the surgeon with 2% lidocaine and 7,5% Ropivacaine. The cumulative dose of anesthetics drugs was computed as not to exceed the recommended dosage.
  To improve patient comfort through the procedure, sedation with Target Controlled Infusion of propofol (using Schnider algorithm) and low dose remifentanil (0,05 mcg/kg/min) was also administered.
  Interventions: Procedure: Regional awake anesthesia
- General anesthesia: Either epidural block or an interfascial plane block of the thoracic wall, such as serratus anterior plane block or erector spinae plane block, were performed.
  Patients were then anesthetized with Propofol plus opiates (usually remifentanil) and muscle paralysis was achieved with Rocuronium.

INTERVENTIONS:
Procedure: Regional awake anesthesia — We want to assess the impact of regional anesthesia on diaphragmatic function in patients undergoing Video-assisted thoracoscopic surgery pulmonary biopsy in interstitial lung disease
  Groups: Regional awake anesthesia

SUMMARY:
Awake thoracic surgery is a feasible and safe alternative to general anesthesia for pulmonary biopsy in interstitial lung disease patients, but there is still no evidence as to its superiority in terms of outcome. However, there is extensive literature about the effect of anesthetic drugs and surgery on diaphragmatic function. Furthermore, in thoracic surgery, diaphragmatic dysfunction was associated with a higher occurrence of postoperative pulmonary complications.

To assess the impact of general anesthesia on diaphragmatic function, the investigators conducted an observational prospective trial. The investigators measured both diaphragmatic excursion and Thickening Fraction at baseline and 12 hours after surgery together with pulmonary function tests and gas exchange data.

DETAILED DESCRIPTION:
Awake thoracic surgery is a feasible and safe alternative to general anesthesia for pulmonary biopsy in interstitial lung disease patients, but there is still no evidence as to its superiority in terms of outcome.

However, there is extensive literature about the effect of anesthetic drugs and surgery on diaphragmatic function. Furthermore, in thoracic surgery, diaphragmatic dysfunction was associated with a higher occurrence of postoperative pulmonary complications.

To assess the impact of general anesthesia on diaphragmatic function, the investigators conducted an observational prospective trial. The investigators measured both diaphragmatic excursion and Thickening Fraction at baseline and 12 hours after surgery together with pulmonary function tests and gas exchange data.

The investigators divided our population into two groups: one group of patients undergoing awake thoracic surgery with epidural anesthesia, and the other group undergoing general anesthesia.

Forty-one patients were recruited and the Thickening Fraction percentage, calculated as (End Inspiratory thickness-End Expiratory thickness)/End Expiratory thickness, was evaluated by means of an ultrasound-assisted method, using a high frequency (10 MHz) linear probe.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for lung biopsy from February 2019 to September 2020

Exclusion Criteria:

* pregnancy,
* Body Mass Index >35,
* Inability to provide informed consent,
* American Society of Anesthesiologists physical status classification score of IV
* Recommended postoperative ICU care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for lung biopsy were enrolled prospectively starting from February 2019 to September 2020.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic maximal function | 12 hours
  Measured with diaphragmatic excursion

SECONDARY OUTCOMES:
Pain scores | 24 hours
  Numeric rate scale
Postoperative Nausea and Vomiting | 24 hours
  Presence/absence of Postoperative Nausea and Vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Luca Brazzi, Professor, Study Chair — University of Torino
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Turin, Italy